CLINICAL TRIAL: NCT01653483
Title: A Randomized, Double-blind, Placebo-controlled, Repeat Dose, 2-period Incomplete Block Crossover Safety and Pharmacokinetic Study of Umeclidinium in Adolescent Asthma Subjects
Brief Title: Aura Adolescent PK Study GSK2829332
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: FDA advised that study is no longer required
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 116213
Record Dates: First submitted 2012-07-23; First posted 2012-07-31 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Asthma
Keywords: Asthma; Umeclidinium; Adolescent; Pharmacokinetics
MeSH Terms: conditions — Asthma | interventions — GSK573719

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK573719 (Experimental): Investigational treatment - Swedish Orange Coloured, opaque hard gelatin capsule
  Interventions: Drug: GSK573719matched-placebo
- GSK573719 matched-placebo (Placebo Comparator): Placebo
  Interventions: Drug: GSK573719

INTERVENTIONS:
Drug: GSK573719 — Novel Dry-Powder Inhaler
  Other Names: umeclidinium
  Arms: GSK573719 matched-placebo
Drug: GSK573719matched-placebo — Novel Dry-Powder Inhaler
  Arms: GSK573719

SUMMARY:
This is a randomized, double-blind, placebo-controlled, repeat dose, 2-period, incomplete block, crossover, safety and pharmacokinetic (PK) study to evaluate 3 once-daily doses of umeclidinium (GSK573719; UMEC) in adolescent asthma subjects aged 12 through 17 years,) who are currently using asthma medications that do not contain inhaled corticosteroids (non-ICS). The objectives are to investigate safety and tolerability, and PK after a 7-day (+2) repeat once-daily dose of UMEC (15.6, 62.5, and 250 mcg) in asthmatic adolescent subjects. Safety endpoints will include reported adverse events, vital signs, ECGs, clinical laboratory tests, and rescue albuterol use. The PK endpoints will include serial PK (plasma and urine) concentrations and derived parameters.

Twenty four subjects will be randomized to participate in the study for up to 7 weeks (including: an initial screening visit, a 7 to 14-day run-in, and 2 treatment periods each of 7 (+2) day duration, with a washout period of 7-14 days between treatment periods). There will be a Follow-up Visit approximately one week after the end of the second treatment period. Subjects will refrain from using rescue medication for 4 hours prior to any clinic visits, unless for emergency.

During each treatment period, study medication will be taken once in the morning until the morning of Day 7 (+2 days) when subjects will return to the clinic for study assessments and take the last dose of study medication. On Day 7 (+2), subjects will remain in the clinic overnight for serial assessments (ECG, and PK plasma and urine samples over the 24-hours).

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, repeat dose, 2-period, incomplete block, crossover, safety and pharmacokinetic (PK) study to evaluate 3 once-daily doses of umeclidinium (UMEC) in adolescent asthma subjects aged 12 through 17 years,) who are currently using asthma medications that do not contain inhaled corticosteroids (non-ICS). The objectives are to investigate safety and tolerability, and PK after a 7-day (+2) repeat once-daily dose of UMEC (15.6, 62.5, and 250 mcg) in asthmatic adolescent subjects. Safety endpoints will include reported adverse events, vital signs, ECGs, clinical laboratory tests, and rescue albuterol use. The PK endpoints will include serial PK (plasma and urine) concentrations and derived parameters.

ELIGIBILITY:
Demographic Inclusion Criteria:

* Informed consent: At least one parent/guardian has signed and dated the written informed consent prior to admission to the study. This will be accompanied by informed assent from the subject for children aged 12 through 17 years.
* Type of Subject: Outpatients. However subjects will remain in the clinic overnight at the end of each treatment period for serial safety and PK blood and urine assessments over a 24-hour period.
* Age: subjects aged 12 through 17 years (inclusive) at Visit 1 (a subject may not participate if the subject's 18th birthday would occur during the conduct of the study). Note: The study population will include an adequate representation of subjects throughout the ages of 12 to 17 years with at least 4 subjects 12 or 13 years of age and no more than 4 subjects 16 or 17 years of age.
* Weight: Subjects must weigh at least 32kg.
* Male or Eligible Female. Eligible being defined as of non-childbearing potential or childbearing potential using an acceptable method of birth control consistently and correctly. Note: To be eligible for entry into the study, females of childbearing potential must commit to consistent and correct use of an acceptable method of birth control, as defined below: Females of childbearing potential who are not sexually active must commit to complete abstinence from intercourse throughout the clinical trial and for a period after the trial to account for elimination of the drug (minimum of 6 days); Male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female subject; Implants of levonorgestrel or etonogestrel; Injectable progestogen; Oral contraceptive (either combined or progestogen alone); Estrogenic vaginal ring; Percutaneous contraceptive patches; Any intrauterine device (IUD) with a documented failure rate of less than 1% per year; Male condom combined with a vaginal spermicide (foam, gel, film, cream, or suppository); Male condom combined with a female diaphragm, either with or without a vaginal spermicide (foam, gel, film, cream, or suppository); Contraceptive transdermal patch, Ortho Evra (if the subject is less than 198 pounds [90kg]); Female subjects should not be enrolled if they are pregnant or lactating or if they plan to become pregnant during the time of study participation. A serum pregnancy test is required of all females and will be performed at the initial screening visit (Visit 1). In addition, a urine pregnancy test will be performed as in the Table of Time and Events.
* Understand protocol requirements: The subject and parent/guardian are able to understand and comply with protocol requirements, instructions, and protocol stated restrictions. The parent or guardian must have the ability to read, write, and record diary information collected throughout the study. The parent or guardian must have the ability to manage study drug administration.

Asthma-Related Diagnostic Inclusion Criteria

* Diagnosis: diagnosis of asthma as defined by the National Institutes of Health [NIH, 2007] at least 6 months prior to Visit 1.
* Severity of Disease: A best pre-bronchodilator AM FEV1 of greater than and equal to 80% of the predicted normal value at the Visit 1 (screening) visit. Percent predicted normal values will be based upon: NHANES III (Hankinson, 1999) for the primary race/ethnicity of the subject (e.g Mexican-American, African-American/African heritage, Caucasian); Multiethnic spirometric assessments (Hankinson, 2010) for the primary race/ethnicity of the subject (e.g Asian).
* Current Anti-Asthma Therapy: Subjects must demonstrate a need for use of a non-corticosteroid medication as shown by having or received a prescription for either of the following for greater than and equal to 12 weeks preceding Visit 1 (and with no ICS used for at least 12 weeks prior to screening): a non-corticosteroid controller (e.g., theophylline, cromolyn, nedocromil, leukotriene modifiers [e.g. montelukast, zafirlukast], etc.), with or without SABA; a SABA bronchodilator such as albuterol.
* Short-Acting Beta2-Agonists (SABAs): All subjects must be able to replace their current SABA treatment with albuterol aerosol inhaler at Visit 1, as needed, for the duration of the study. Subjects must be judged capable of withholding albuterol for at least 4 hours prior to study visits.

Demographic Exclusion Criteria

* Tobacco Use: A subject may not have used inhaled tobacco products (i.e., cigarettes, cigars, or pipe tobacco) or have historical use of tobacco products. Includes, urinary cotinine or CO breath test levels at screening that is indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Previous Use of Study Drug or Investigational Products: Previous use of UMEC excludes a subject or the subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Compliance: A subject will not be eligible if he/she or his/her parent or legal guardian has any infirmity, disability, disease, or geographical location which seems likely (in the opinion of the investigator) to impair compliance with any aspect of this study protocol, including visit schedule and completion of the daily diaries.
* Alcohol or substance abuse: Subjects with any history of alcohol use or substance abuse prior to screening, or use of, at any time during the study.
* Viral Hepatitis: A positive Hepatitis B surface antigen or positive Hepatitis C antibody pre-study or at Visit 1.
* Wards of State: Children who are wards of the state or government.
* Affiliation with Investigator's Site: A subject will not be eligible for this study if he/she is an immediate family member of the participating investigator, sub-investigator, study coordinator, or employee of the participating investigator.
* Pregnancy: Pregnant females as determined by positive serum hCG test at screening or prior to dosing.
* Lactation: Lactating females.

Asthma-Related Exclusion Criteria

* History of Life-threatening asthma: Defined for this protocol as an asthma episode that required intubation and/or was associated with hypercapnea requiring non-invasive ventilator support, respiratory arrest, hypoxic seizures or asthma-related syncopal episode(s).
* Asthma Exacerbation: A subject must not have a history of a severe asthma exacerbation within 12 weeks prior to Visit 1. A severe asthma exacerbation is defined as deterioration of asthma requiring the use of systemic corticosteroids (oral, or injection) for at least 3 days or an inpatient hospitalization or emergency department visit due to asthma that required systemic corticosteroids.
* Signs or symptoms of unstable asthma: Defined as: During the 7 days immediately preceding a visit, at least 3 days in which greater than and equal to 12 inhalations/day of albuterol/salbutamol were used; or A symptom score of greater than and equal to 4 on at least 3 consecutive days during the previous 7 days (defined as the subject experiencing symptoms for most of the day which affected normal daily activities); or at the discretion of the Investigator
* Respiratory Infection expected to affect the subject's ability to participate in the study: Within 4 weeks prior to Visit 1 a subject has had a culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus or middle ear that is not resolved and has led to a change in asthma management or, in the opinion of the Investigator, is expected to affect the subject's asthma status or the subject's ability to participate in the study.
* Concurrent Respiratory Disease: A subject must not have current evidence of pneumonia, pneumothorax, atelectasis, pulmonary fibrotic disease, bronchopulmonary dysplasia, chronic bronchitis, emphysema, chronic obstructive pulmonary disease, or other respiratory abnormalities other than asthma.
* Diseases Preventing Use of Anticholinergics: Diagnosis of narrow-angle glaucoma, or bladder neck obstruction that in the opinion of the study investigator or GSK medical monitor would pose a safety risk with use of an inhaled anticholinergic.
* Other Concurrent Diseases/Abnormalities: A subject must not have any clinically significant, uncontrolled condition or disease state that, in the opinion of the investigator, would put the safety of the patient at risk through study participation if the condition/disease exacerbated during the study. The investigator is encouraged to contact the study medical monitor if further clarification is warranted.

Safety Exclusion Criteria

* Liver Function: ALT greater than and equal to 2xULN; alkaline phosphatase and bilirubin greater than and equal to 1.5xULN (isolated bilirubin less than 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin less than 35%).
* Average QTcF greater than 450 msec.
* Allergies: Drug Allergy - Any adverse reaction including immediate or delayed hypersensitivity to any beta-agonist, or sympathomimetic drug. Known or suspected sensitivity to the constituents of the NDPI (i.e., lactose).
* Previous Clinical Trials: Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Concomitant Medication or Treatments: Administration of prescription or over-the-counter medication that would significantly affect the course of asthma, or interact with study drug, such as:: Medication: Mucolytics such as acetylcysteine; beta -blocker eye drops ( e.g. use in glaucoma symptoms treatment) or systemic beta-adrenergic blocking agents; No use within the following time interval before Visit 1: 12 weeks. Medication: Inhaled short-acting beta2-agonists (rescue use albuterol is permitted during the study); No use within the following time interval before Visit 1: 4 hours (including all study visits). Medication: Short acting anticholinergics; No use within the following time interval before Visit 1: 6 hours. Medication: Long and short acting oral beta2-agonists; No use within the following time interval before Visit 1: 24 hours. Medication: Long acting anticholinergics or antimuscarinics; No use within the following time interval before Visit 1: 14 days. Medication: Systemic, depot, or oral corticosteroids; No use within the following time interval before Visit 1: 4 weeks. Medication: Inhaled corticosteroids (ICS); No use within the following time interval before Visit 1: 12 weeks. Medication: Inhaled long-acting beta2-agonists (e.g. salmeterol, formoterol, indacaterol) including long-acting beta2-agonists combined with an ICS (e.g. Advair, seretide); No use within the following time interval before Visit 1: 4 weeks. Medication: Immunosuppressive medications (e.g., methotrexate, gold, or dapsone) including immunomodulators (Immunotherapy for the treatment of allergies is allowed during the study provided it was initiated at least 4 weeks prior to Visit 1 and the subject remains in the maintenance phase throughout the study); No use within the following time interval before Visit 1: 12 weeks. Medication: Monoclonal antibody: Anti-IgE, or any other monoclonal antibody, for any reason (e.g., omalizumab); No use within the following time interval before Visit 1: 5 months. Medication: Strong and moderate pgp inhibitors (e.g. dronedarone,ritonavir, indinavir, quinidine, valspodar, elacridar (GF120918); No use within the following time interval before Visit 1: 4 weeks. Medication: Strong and moderate CYP2D6 inhibitors (bupropion, fluoxetine, paroxetine, quinidine, ecstasy, terbinafine, cinacalcet, ritonavir, tipranavir, moclobemide, duloxetine, dronedarone); No use within the following time interval before Visit 1: 4 weeks. Medication: Any other investigational drug; No use within the following time interval before Visit 1: 30 days or within 5 drug half-lives of the investigational drug (whichever is longer) - Liver Disease: Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Bundle branch block: Subjects with right or left bundle branch block.
* Blood Volume: Where participation in the study would result in donation of blood or blood products in excess of 500mL within a 56-day period.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2012-09 (Actual); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Subject safety as measured by serial ECGs and vital signs measured on Days 7 of each treatment period and the number (and frequency) of subjects who experience adverse events after repeat doses of GSK573719 | Through the expected 7 day duration for each of 2 treatment periods.
  Assessment of safety and tolerability, including: reported adverse events, clinical laboratory measurements, vital signs (heart rate and blood pressure), and electrocardiographic (ECG) parameters.

SECONDARY OUTCOMES:
Subject safety as measured by ECGs and vital signs measures on Day 1 of each treatment period | Through the expected 6 hour duration of in clinic stay
  Assessment of safety and tolerability, including: vital signs (heart rate and blood pressure), and electrocardiographic (ECG) parameters.
Pharmacokinetic parameters such as Cmax, AUC, half-life, Tmax of GSK573719 after repeat dosing. | predose, 5, 15 and 30 minutes and, 1, 2, 4, 6, 8, 12, and 24, hours on Day 7 of dosing
  To characterise the PK profile of repeat doses of GSK573719 in adolescent asthmatic subjects

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline